CLINICAL TRIAL: NCT01279538
Title: A Phase 1b, Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Single-Dose, Pharmacokinetic, Pharmacodynamic, Safety and Tolerability Study of ASKP1240 in de Novo Kidney Transplantation
Brief Title: A Study to Assess Pharmacokinetic, Pharmacodynamic, Safety and Tolerability of ASKP1240 in de Novo Kidney Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7163-CL-0103
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation
Keywords: Pharmacology; Pharmacokinetics; ASKP1240; Kidney Transplantation
MeSH Terms: interventions — bleselumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ASKP1240 lowest dose (Experimental): Participants received a single 30-minute study drug infusion on Study Day 1, followed by a 90-day follow-up period.
  Interventions: Drug: bleselumab
- ASKP1240 low dose (Experimental): Participants received a single 30-minute study drug infusion on Study Day 1, followed by a 90-day follow-up period.
  Interventions: Drug: bleselumab
- ASKP1240 high dose (Experimental): Participants received a single 30-minute study drug infusion on Study Day 1, followed by a 90-day follow-up period.
  Interventions: Drug: bleselumab
- ASKP1240 highest dose (Experimental): Participants received a single 30-minute study drug infusion on Study Day 1, followed by a 90-day follow-up period.
  Interventions: Drug: bleselumab
- Placebo (Placebo Comparator): Participants received a single 30-minute matching placebo infusion on Study Day 1, followed by a 90-day follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bleselumab — Intravenous (IV) infusion
  Other Names: ASKP1240
  Arms: ASKP1240 high dose; ASKP1240 highest dose; ASKP1240 low dose; ASKP1240 lowest dose
Drug: Placebo — Intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the Pharmacokinetics (PK),

pharmacodynamics (PD), safety and tolerability of ASKP1240 when administered to subjects who received a de novo kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a recipient of a de novo kidney transplant from a living or deceased donor
* Prior to randomization, the subject has a post-transplant serum creatinine value that is at least 30% decreased from the pre-transplant value and requires no dialysis
* Female subject of child bearing potential must have a negative serum pregnancy test within 7 days prior to enrollment or upon hospitalization and must agree to maintain effective birth control during the study
* All sexually active male subjects must agree to use an adequate method of contraception throughout the study period and for 90 days after the last dose of study drug and agrees to no sperm donation until the end of the study, or for 90 days after the last dose of study drug, whichever is longer
* Subject must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions

Exclusion Criteria:

* Prior to randomization, subject will receive antibody induction therapy (e.g., thymoglobulin, basiliximab, daclizumab, OKT3, alemtuzumab)
* Subject has previously received or is receiving an organ transplant other than a kidney
* Recipient has a positive T or B cell crossmatch
* Subject has ABO blood type incompatibility with their donor
* Subject has received intravenous immunoglobulin (IVIG) therapy in the 3 months prior to first dose of study drug
* Recipient or donor is known by medical history to be seropositive for human immunodeficiency virus (HIV)
* Subject had a thromboembolic event (e.g., myocardial infarction, cerebrovascular event, pulmonary embolus, deep vein thrombosis, peripheral arterial thromboembolic event) in the past 5 years or if the subject is on specific therapy for prophylaxis or treatment of such an event. Low dose aspirin (81 mg) therapy is not considered exclusionary. NOTE: A one-time event of arterio-venous (AV) fistula dialysis access thrombosis is not exclusionary. Subjects with recurrent AV fistula thrombosis or those on systemic medications to prevent reoccurrence are excluded
* Subject has a current malignancy or a history of any malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Subject has an uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives
* Subject is concurrently participating in another drug study or has received an investigational drug up to 8 weeks (depending on medication) prior to transplant
* Subject has previously received ASKP1240 or participated in a study involving ASKP1240
* Subject has abnormal chest x-ray indicative of acute or chronic lung disease on a prior examination within 3 months prior to randomization
* Subject has abnormal electrocardiogram (ECG) considered as clinically significant on a prior examination within 3 months prior to randomization
* Subject has uncontrolled intercurrent illness, including, but not limited to ongoing or active infection, any clinically significant cardiac disease, seizure disorder, or psychiatric illness/social situations that would limit compliance with study requirements
* Subject has received live or live attenuated virus vaccinations within the last 30 days prior to first dose of study drug
* Subject has a clinical condition which would not allow safe conduct and completion of the study
* Subject is pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11-17 (Actual); Primary Completion 2012-01-23 (Actual); Study Completion 2012-01-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment through analysis of blood samples | Up to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (21):
- United States (21):
  - Stanford University Medical Center, Palo Alto, California
  - California Institute of Renal Research, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Illinois Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, The Transplant Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Barnabas Medical Center, Livingston, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati - University Internal Medicine Associates, Cincinnati, Ohio
  - Central Pennsylvania Transplant Associates, Harrisburg, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency.

REFERENCES:
- [Derived] Vincenti F, Klintmalm G, Yang H, Ram Peddi V, Blahunka P, Conkle A, Santos V, Holman J. A randomized, phase 1b study of the pharmacokinetics, pharmacodynamics, safety, and tolerability of bleselumab, a fully human, anti-CD40 monoclonal antibody, in kidney transplantation. Am J Transplant. 2020 Jan;20(1):172-180. doi: 10.1111/ajt.15560. Epub 2019 Sep 9. PMID 31397943
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/7163-CL-0103/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25562&tenant=MT_AST_9011